CLINICAL TRIAL: NCT05286463
Title: Effect of Ultrasound-enhanced Bee Venom on Selected Post Inguinal Hernioplasty Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohamed othman, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: /012/002764
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Complications; C, Intestinal (Internal)
Keywords: phonophoresis, inguinal hernioplasty, bee venom

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): received low-intensity pulsed ultrasound using bee venom (BV) gel for 5 minutes for each session, three times a week, for three consecutive weeks postoperative and received regular medical care.
  Interventions: Combination Product: bee venom gel phonophoresis
- group B (Sham Comparator): received low-intensity pulsed ultrasound using only plain gel without BV gel for 5 minutes for each session, three times a week, for three consecutive weeks postoperative and received regular medical care.
  Interventions: Device: low intensity ultrasound

INTERVENTIONS:
Combination Product: bee venom gel phonophoresis — a noncontact low-frequency pulsed ultrasound delivered through Bee Venom previously prepared gel as topical application using an ultrasonic therapy instrument with frequency, 0.5-MHZ pulsed mode (applicator 1.9 cm2) applied around the incision site, Ren 4 and Ren 6. The movement was over the incision margins, Ren 4 and Ren 6 with a pulsed duty cycle of 40% (4 ms on, 6 ms off), and power density of 0.5 W/cm2, Before and after each patient exposure, the ultrasonic applicator's performance was tested on a regular basis, and each test included all essential acoustic field characteristics (pressure amplitude, frequency), as well as the uniformity of the field distribution.
  Other Names: low intensity Ultrasound with bee venom gel
  Arms: group A
Device: low intensity ultrasound — a noncontact low-frequency pulsed ultrasound delivered through plain gel only using an ultrasonic therapy instrument with frequency, 0.5-MHZ pulsed mode (applicator 1.9 cm2) applied around the incision site, Ren 4 and Ren 6. The movement was over the incision margins, Ren 4 and Ren 6 with a pulsed duty cycle of 40% (4 ms on, 6 ms off), and power density of 0.5 W/cm2, Before and after each patient exposure, the ultrasonic applicator's performance was tested on a regular basis, and each test included all essential acoustic field characteristics (pressure amplitude, frequency), as well as the uniformity of the field distribution.
  Arms: group B

SUMMARY:
Objectives: Bee venom phonophoresis has been suggested as a noninvasive treatment for a number of inflammatory conditions and to reduce postoperative pain. The aim of this study was to evaluate the effect of bee venom phonophoresis on selected acupuncture points for the treatment of pain, inflammation, and mobility of the hip following inguinal hernioplasty.

HYPOTHESES:

It will be hypothesized that:

It was hypothesized that Bee venom phonophoresis has no or limited effect in improvement of post inguinal hernioplasty complication.

RESEARCH QUESTION: Does Bee venom phonophoresis an effect in improvement of post inguinal hernioplasty complication?

DETAILED DESCRIPTION:
All patients in both groups of the study (A) and (B) would receive a noncontact low-frequency pulsed ultrasound delivered through a fine mist of sterile saline or alcohol at the incisional site of inguinal hernioplasty, REN 4 and REN 6. Treatment sessions were 3 sessions a week for 3 consecutive weeks. Before and after each patient exposure, the ultrasonic applicator's performance was tested on a regular basis, and each test included all essential acoustic field characteristics (pressure amplitude, frequency), as well as the uniformity of the field distribution.

Ren 4: On the anterior midline, 2 sun superior to the upper border of the pubic symphysis or 3 sun inferior to the umbilicus. Ren 6: On the anterior midline, 1.5 sun inferior to the umbilicus or 3.5 sun superior to the upper border of the pubic symphysis.

For the bee venom phonophoresis group (A): A single clinical dosage of diluted bee venom (BV) in normal saline, 0.05 ml (1 g/ml), was injected into the forearm via either an intradermal or subcutaneous method to test for BV allergy. Subjects might take part in this study if the examined lesion caused a wheal with a diameter of less than 10 mm and an erythema with a diameter of less than 26.5 mm after 10 to 15 minutes.28 Participants were treated with BV previously prepared gel as topical application using an ultrasonic therapy instrument with frequency, 0.5-megahertz pulsed mode (applicator 1.9 cm2) applied around the incision site. The movement was over the incision margins with a pulsed duty cycle of 40% (4 ms on, 6 ms off), and power density of 0.5 W/cm2, and time was 5 minutes each session. Each participant was put in the most comfortable and relaxed position as a supine lying position, and the patient was asked to expose the incision site to avoid any restriction for receiving phonophoresis around the incisional site, REN 4 and REN 6. The incision margin was cleaned with alcohol or normal saline, the ultrasound unit's plug was inserted into the main current supply, and the treatment approach (phonophoresis application for bee venom gel) was prepared; each participant received a total amount of about 0.6 mg to 1 mg of BV gel each session for a total of 5 minutes.29 The participants in the control group (Group B) received only low-intensity pulsed ultrasound applied around the incisional site, REN 4 and REN 6 for 5 minutes, as in Group A, using only plain gel without BV gel.

ELIGIBILITY:
Inclusion Criteria:

* Patients ranged in age from 28 to 50 years old.
* They had not previously undertaken another physical therapy modality for pain
* Non-smokers
* Under their own prescribed medications described by their physicians.

Exclusion Criteria: Patients were excluded if they:

* had non-mesh inguinal hernioplasty.
* suffered from open or infected wounds.
* had any systemic diseases that may interfere with the study's objectives such as using chemo or radiotherapy.
* had allergy to bee venom.
* had associated disorders, such as immunodeficiency, HIV, diabetes, or anemia.

Ages: 28 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Serum C-reactive protein (CRP) | change in CRP calculated at post-3 weeks of treatment minus baseline.
  blood sample analyzed at laboratory unit
Manual Goniometer | change in ranges of motion calculated at post-3 weeks of treatment minus baseline.
  A simple long-arm goniometer with a 360° scale marked in one-degree increments was used. A manual goniometer was used for assessment of hip flexion, extension, abduction, and adduction range of motion (ROM).
The visual analogue scale (VAS) | change in VAS calculated at post-3 weeks of treatment minus baseline.
  The visual analogue scale (VAS) is a 10-cm-long line with the ends labelled as the pain extremes (e.g., no pain to unbearable pain). Between "no pain" and "worst pain," patients were asked to mark the spot on the line that best described their pain experience. The operator then measured in millimetres the gap between zero and "no pain".

CONTACTS AND LOCATIONS:
Overall Officials: eman othman, professor, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in bee venom or ulcer . we will share the results of this study within 1 year following publication
Supporting Information: SAP, ICF
Time Frame: within 1 year following publication
Access Criteria: the criteria will be assessed by the publication of the trial in an international journals.